CLINICAL TRIAL: NCT00551512
Title: Phase I Clinical and Pharmacokinetic Study of CBP501 and Cisplatin Every 3 Weeks in Patients With Advanced Refractory Solid Tumors
Brief Title: Phase I Study of CBP501 and Cisplatin in Patients With Advanced Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CanBas Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBP 06-01
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Cancer; Solid Tumors
Keywords: cancer; solid tumors
MeSH Terms: conditions — Neoplasms | interventions — Cdc25C phosphatase (211-221); Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CBP501 and Cisplatin (Experimental): Dose escalation study
  Interventions: Drug: CBP501 and Cisplatin

INTERVENTIONS:
Drug: CBP501 and Cisplatin — CBP501 is given IV on Day 1 of each cycle (every 21 days). Dose escalation of CBP501 and cisplatin will be starting doses of 3.6 mg/m² CBP501 and 50 mg/m² cisplatin (Dose Level 1). Step 1, if during the first 2 cycles, at least 2 out of 3 to 6 patients experience Dose Limiting Toxicity (DLT) at 50 mg/m² cisplatin, then the cisplatin dose will be de-escalated to 30 mg/m². If no more than 1 out of 6 patients experiences DLT, cisplatin dose will be escalated to 75 mg/m². Step 2, dose escalation will be performed using the cisplatin MTD, with escalating CBP501 doses. CBP501 dose escalation will take place until the MTD has been defined or 74 mg/m² is reached.
  Other Names: CBP501 and CDDP

SUMMARY:
The purpose of this research study is to find the answers to the following questions:

1. What are the highest doses of CBP501 and cisplatin that can be safely administered as consecutive 2-hours and 1-hour infusions every 21 days?
2. What are the side effects of the combination of CBP501 and cisplatin when given as an infusion every 21 days?
3. What amount of CBP501 and cisplatin are found in the blood at certain times after it is given?
4. Are there any substances in your blood or tumor that can tell us about tumor sensitivity to CBP501 and cisplatin?
5. Will CBP501 given with cisplatin help to treat your cancer?

DETAILED DESCRIPTION:
9.1 23BOverall Study Design and Plan This was an open-label, multicenter, dose-escalation and pharmacokinetic Phase I study of CBP501 and cisplatin administered as consecutive IV infusions according to a once-every-3-weeks schedule in patients with advanced solid tumors refractory to standard therapy. The study was conducted in three US centers. During the course of the study, an amendment was introduced (#3, October 17th, 2007; see section X9.8X) to allow administration of a unique dosing of single agent CBP501 prior to the initiation of combination therapy to enable completion of the pharmacokinetic (PK) characterization of single agent CBP501. Pharmacodynamic analysis involving phosphoserine 216 evaluations was also removed. See section X16.1.1X for copies of the protocol and all protocol amendments. With 8 additional patients included at the recommended dose (at DL6), it was decided to stop all PK and CTC sampling (and therefore the day-7 CBP501 alone infusion), as sufficient information had been retrieved. In addition, based on evidence of efficacy observed in ovarian cancer patients, a further 10 ovarian and 4 endometrial cancer patients were to be included at the recommended dose; these patients were to be assessed for DLT to confirm the identification of the MTD.

Case Report Forms were used to collect the data, and data management was carried out by AAIOncology. All laboratory data and Investigator observations were be transcribed into the CRF. ECG, U/S, MRI and CT scans were to be reported in summary in the CRF. The original reports, traces and films were to be retained by the Investigators for future reference. See section X16.1.2X for a sample CRF.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to initiation of any study-specific procedures.
* Pathologically-confirmed, locally advanced or metastatic solid tumors, refractory to standard therapy.
* Male or female patients aged 18 years or over.
* ECOG Performance Status (PS): 0-1.
* Life expectancy > 3 months.
* Previous anticancer treatment must be discontinued at least 3 weeks prior to first dose of study treatment (6 weeks for mitomycin C; 6 weeks for anti-androgen therapy if discontinued prior to treatment initiation, with the exception of 8 weeks for bicalutamide).
* Adequate organ function including the following:
* Bone Marrow: absolute neutrophil count (ANC) ³ 1.5 x 109/L, platelet count ³ 100 x 109/L, hemoglobin ³ 9 g/dL
* Hepatic: Bilirubin £ 1.5 x the upper limit of normal (ULN), aspartate transaminases (AST/SGOT) and alanine transaminases (ALT/SGPT) £ 2.5 x ULN (or ≤ 5 x ULN if liver metastases are present), INR £ 1.5 x ULN
* Renal: Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ³ 70 mL/min (calculated according to the Cockroft and Gault formula)
* Metabolic: serum potassium, calcium and magnesium ³ lower limit of normal (LLN)
* Creatine phosphokinase isoenzymes: CPK-MB, CPK-MM ≤ ULN
* Troponin I serum level within normal values
* Female patients of child-bearing potential must have a negative pregnancy test and use at least one form of contraception as approved by the investigator for 4 weeks prior to the study and 4 months after the last dose of study drug. For the purposes of this study, child-bearing potential is defined as: "All female patients unless they are post-menopausal for at least one year or are surgically sterile".
* Male patients must use a form of barrier contraception approved by the investigator during the study and for 4 months after the last dose of study drug.
* Ability to co-operate with the treatment and follow-up.

Exclusion Criteria:

* Radiation therapy to more than 30% of the bone marrow prior to entry into the study.
* Prior chemotherapy with nitrosoureas or high dose carboplatin (AUC > 6 mg/mL), prior mitomycin C cumulative dose ³ 25 mg/m², prior bone marrow transplant or intensive chemotherapy with stem cell support.
* Presence of any serious concomitant systemic disorders incompatible with the study (e.g. uncontrolled congestive heart failure, active infection, etc.).
* Any previous history of another malignancy (other than cured basal cell carcinoma of the skin or cured in-situ carcinoma of the cervix) within 5 years of study entry.
* Presence of any significant central nervous system or psychiatric disorder(s) that would hamper the patient's compliance.
* Evidence of peripheral neuropathy > grade 1 according to NCI-CTCAE Version 3.
* Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to study entry.
* Pregnant or breast-feeding patients or any patient with childbearing potential not using adequate contraception.
* Known HIV, HBV, HCV infection.
* Active CNS metastasis: patients with a history of CNS metastases will be eligible if they have been treated and are stable without symptoms for 4 weeks after completion of treatment, with image documentation required, and must be either off steroids or on a stable dose of steroids for > 1 week prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) during the first two treatment cycles | 6 weeks

SECONDARY OUTCOMES:
Incidence and severity of adverse events and laboratory abnormalities, graded according to NCI-CTCAE version 3.0 | During and at end of study
Occurrence of Serious Adverse Events (SAEs) | During and at end of study
Occurrence of discontinuations due to treatment-related adverse events | At end of study
Serum concentrations of CBP501 and total and ultrafiltrate platinum to determine, via non-compartmental methods, Cmax, AUC, lz, t½, Cl and Vss. | During and at end of study
Evaluation of the relationship between administered dose and plasma pharmacokinetic parameters for CBP501 and cisplatin | During and at end of study
Objective tumor response assessed according to RECIST | During and at end of study
Time to progression | During and at end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Wasserman, MD, Study Director — AAIOncology
Locations (3):
- United States (3):
  - Scottsdale Clinical Research Institute, Scottsdale, Arizona
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Nevada Cancer Institute, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mine N, Yamamoto S, Saito N, Yamazaki S, Suda C, Ishigaki M, Kufe DW, Von Hoff DD, Kawabe T. CBP501-calmodulin binding contributes to sensitizing tumor cells to cisplatin and bleomycin. Mol Cancer Ther. 2011 Oct;10(10):1929-38. doi: 10.1158/1535-7163.MCT-10-1139. Epub 2011 Aug 10. PMID 21831962
- [Background] Sha SK, Sato T, Kobayashi H, Ishigaki M, Yamamoto S, Sato H, Takada A, Nakajyo S, Mochizuki Y, Friedman JM, Cheng FC, Okura T, Kimura R, Kufe DW, Vonhoff DD, Kawabe T. Cell cycle phenotype-based optimization of G2-abrogating peptides yields CBP501 with a unique mechanism of action at the G2 checkpoint. Mol Cancer Ther. 2007 Jan;6(1):147-53. doi: 10.1158/1535-7163.MCT-06-0371. PMID 17237275
- [Background] Suganuma M, Kawabe T, Hori H, Funabiki T, Okamoto T. Sensitization of cancer cells to DNA damage-induced cell death by specific cell cycle G2 checkpoint abrogation. Cancer Res. 1999 Dec 1;59(23):5887-91. PMID 10606229
- [Background] Matsumoto Y, Shindo Y, Takakusagi Y, Takakusagi K, Tsukuda S, Kusayanagi T, Sato H, Kawabe T, Sugawara F, Sakaguchi K. Screening of a library of T7 phage-displayed peptides identifies alphaC helix in 14-3-3 protein as a CBP501-binding site. Bioorg Med Chem. 2011 Dec 1;19(23):7049-56. doi: 10.1016/j.bmc.2011.10.004. Epub 2011 Oct 7. PMID 22032894
- [Result] Shapiro GI, Tibes R, Gordon MS, Wong BY, Eder JP, Borad MJ, Mendelson DS, Vogelzang NJ, Bastos BR, Weiss GJ, Fernandez C, Sutherland W, Sato H, Pierceall WE, Weaver D, Slough S, Wasserman E, Kufe DW, Von Hoff D, Kawabe T, Sharma S. Phase I studies of CBP501, a G2 checkpoint abrogator, as monotherapy and in combination with cisplatin in patients with advanced solid tumors. Clin Cancer Res. 2011 May 15;17(10):3431-42. doi: 10.1158/1078-0432.CCR-10-2345. Epub 2011 Jan 10. PMID 21220472